CLINICAL TRIAL: NCT00004755
Title: Phase II Randomized Study of Allopurinol Versus Glucantime Versus Allopurinol/Glucantime for Cutaneous Leishmaniasis in Brazil
Brief Title: Allopurinol, Glucantime, or Allopurinol/Glucantime for Cutaneous Leishmaniasis in Brazil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 199/11679; HSPH-11679
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-01

CONDITIONS: Leishmaniasis
Keywords: dermatologic disorders; environmental/toxic disorders; immunologic disorders and infectious disorders; leishmaniasis; rare disease
MeSH Terms: conditions — Leishmaniasis; Skin Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Allopurinol; Meglumine Antimoniate

INTERVENTIONS:
Drug: allopurinol
Drug: glucantime

SUMMARY:
OBJECTIVE:

Compare the efficacy and side effects of allopurinol versus glucantime versus allopurinol/glucantime in patients in Brazil with cutaneous leishmaniasis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized study. Patients are stratified by participating institution.

One group is treated with daily intramuscular injections of glucantime. Patients with less than a complete response on Day 21 continue treatment until lesions heal completely or for a maximum of 60 days. Patients with progressive disease on Day 40 are removed from study.

The second group is treated with daily oral allopurinol. Patients with a partial response on Day 21 continue treatment until lesions heal completely. Patients with stable or progressive disease on Day 21 or unhealed lesions on Day 56 cross to glucantime therapy. Accrual into this group was closed in 6/96.

The third group receives allopurinol and glucantime.

Patients are followed at 3, 6, and 9 months, then annually for at least 5 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Parasitologically confirmed cutaneous leishmaniasis (lesion of less than 3 months duration)

No mucocutaneous leishmaniasis

No prior leishmaniasis

--Prior/Concurrent Therapy--

No prior treatment for leishmaniasis

--Patient Characteristics--

Hepatic: No clinical or laboratory evidence of hepatic disease

Renal: No clinical or laboratory evidence of renal disease No hyperuricemia or gout

Cardiovascular: No clinical, electrocardiographic, or laboratory evidence of cardiac disease

Other: No allergy or other contraindication to allopurinol or glucantime; No concurrent medication that might interact with study drugs, e.g.: probenecid, warfarin, azathioprine; No skin rash; No malnutrition; No other medical contraindication to protocol therapy; No pregnant or nursing women

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 375
Dates: Start 1995-09

CONTACTS AND LOCATIONS:
Overall Officials: James H. Maguire, Study Chair — Harvard School of Public Health (HSPH)